CLINICAL TRIAL: NCT00844935
Title: The Value of Electrocardiographic Autonomic Nervous System Function Measures for Predicting Cardiopulmonary Recovery of Mechanically Ventilated Patients in Intensive Care
Brief Title: Electrocardiographic Autonomic Function Measures in Mechanically Ventilated Patients
Status: Withdrawn | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H6052-33761-01
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Disorders of the Autonomic Nervous System; Cardiovascular Abnormalities; Respiratory Disorders
Keywords: Heart rate variability, mechanical ventilation, weaning,; spontaneous breathing trial
MeSH Terms: conditions — Autonomic Nervous System Diseases; Cardiovascular Abnormalities; Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
This research proposal has two main objectives. The first is to increase understanding of the underlying physiological interactions that occur between the cardiovascular, pulmonary, and ANS during transition between positive pressure mechanical ventilation (MV) and spontaneous breathing. The second is to determine if heart rate variability, (HRV) a reflection of autonomic nervous system (ANS) activity, and autonomic information flow (AIF), a set of nonlinear measures derived from HRV, both measured in the intensive care unit (ICU) can predict patient outcomes including successful weaning and in-hospital recovery time after an episode of cardiopulmonary compromise requiring MV.

Hypothesis 1. Transitions between mechanically supported ventilation and spontaneous breathing will disturb cardiovascular synchrony, altering the relationship of HRV, AIF, respiratory rate, and blood pressure;

Hypothesis 2. More normal HRV and AIF values, measured during baseline MV and sedation awakening (a period immediately prior to SBT when sedative medications are discontinued) will be associated with easier weaning, and shorter intensive care unit (ICU) and hospital lengths of stay; more abnormal measurements will be associated with longer lengths of stay;

Hypothesis 3. AIF is a more sensitive predictor of successful weaning from MV than HRV.

ELIGIBILITY:
Inclusion Criteria:

* Receiving mechanical ventilation in medical-surgical intensive care unit;
* Eighteen years of age or older;
* Expectation of receiving initial spontaneous breathing trial within the next 24 hours.

Exclusion Criteria:

* Pregnant;
* Expectation of non-survival when ventilator is discontinued;
* Cardiac rhythm of atrial fibrillation;
* Paced cardiac rhythm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients in intensive care
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Drew, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco Medical Center, San Francisco, California, United States